CLINICAL TRIAL: NCT05219084
Title: Hip Denervation and Intra-articular Hydration in Damaged Hip in Axial Spondyloarthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC 250
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Patients With Axial SpA According to ASAS Criteria; Patients With Unilateral or Bilater Hip Damage According to BASRI Score; Age > 18
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo group (Placebo Comparator): 5ml of normal; saline-injected subcutaneously
  Interventions: Drug: Control group
- Hip denervatiopn (Active Comparator): Hip denervation with lidocaine 2% to each genicular branch, 2ml at each point
  Interventions: Drug: hip denervation
- Inra-articular hydration (Active Comparator): 10 ml of normal saline injected inside the hip under ultrasound guidance
  Interventions: Drug: intra-articular hydration
- compined group (Active Comparator): hip denervation and intra-articular hydration were conducted together in this group
  Interventions: Drug: Combined group

INTERVENTIONS:
Drug: hip denervation — Lidocaine 2% 2ml was injected into each genicular nerve
  Arms: Hip denervatiopn
Drug: intra-articular hydration — 10 ml; of normal; saline were injected inside the hip joint
  Arms: Inra-articular hydration
Drug: Combined group — hip denervation and intra-articular hydration were conducted together
  Arms: compined group
Drug: Control group — Normal; saline was injected subcutaneously
  Arms: placebo group

SUMMARY:
Background: The hip joint is frequently affected in axial spondyloarthritis (SpA) of adults with destructive effects in untreated patients. About 35% of axial SpA patients had either unilateral or bilateral hip arthritis. Destruction is more common with early-onset, active disease, or enthesitis.

Objectives: The aim of this study is to evaluate the effect of hip denervation (HD) and intra-articular hydration (IAH) on pain, function score, hip mobility scores in a cohort of axial SpA patients with grade 3 and 4 hip BASRI scores.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or more
* Axial; SpA fulfilled ASA criteria
* BASRI score grade 3 or 4 for one hip at least

Exclusion Criteria:

* patients younger than 18
* Axial; SpA with normal hip or hip involvement less than 3 on BASRI score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale | Baseline , after 4 weeks and after 12 weeks
  0 means no pain, 100 means the highest degree of pain
Change in Harris functional hip score | Baseline, after 4 weeks and after 12 weeks
  Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points).
  The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result
Change in range of motion of the hip | Baseline, after 4 weeks and after 12 weeks
  hip flexion, extension , internal; rotation , external; rotation , abduction , and adduction all were recopreded
Change in semiquantitative tenderness score | Baseline, after 4 weeks and after 12 weeks
  a score from 0-3, 90 means no tenderness and 3 means maximum tenderness

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Elsaman, Sohag, Egypt